CLINICAL TRIAL: NCT02298725
Title: Individual Metabolism and Physiology Signature Study
Acronym: iMAPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Collaborators: Dairy Research Institute (Other); University of California, Davis (Other); University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 648620
Record Dates: First submitted 2014-11-18; First posted 2014-11-24 (Estimated); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Insulin Resistance; Metabolic Syndrome X; Obesity
Keywords: Insulin Resistance; Obesity; US Dietary Guidelines
MeSH Terms: conditions — Insulin Resistance; Metabolic Syndrome; Obesity | interventions — Nutrition Policy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- DGA Diet Plan (Experimental): A nutrient-adequate, balanced diet providing energy to maintain body weight, and macronutrient composition falling within the acceptable range, as recommended by the Institute of Medicine. The foods provided in this diet will be closely aligned with food group recommendations set in the 2010 Dietary Guidelines for Americans. All foods and beverages will be provided to enrolled subjects during the intervention period.
  Interventions: Other: DGA Diet Plan
- NHANES Diet Plan (Experimental): A nutrient-adequate, balanced diet providing energy to maintain body weight, and macronutrient composition falling within the acceptable range, as recommended by the Institute of Medicine. The foods provided in this diet plan will be closely aligned with the NHANES "What We Eat In America" report. All foods and beverages will be provided to enrolled subjects during the intervention period.
  Interventions: Other: NHANES Diet Plan

INTERVENTIONS:
Other: DGA Diet Plan — A nutrient-adequate, balanced diet providing energy to maintain body weight, and macronutrient composition falling within the acceptable range, as recommended by the Institute of Medicine. The foods provided in this diet will be closely aligned with food group recommendations set in the 2010 Dietary Guidelines for Americans.
  Other Names: Dietary Guidelines for Americans Diet Plan
  Arms: DGA Diet Plan
Other: NHANES Diet Plan — A nutrient-adequate, balanced diet providing energy to maintain body weight, and macronutrient composition falling within the acceptable range, as recommended by the Institute of Medicine. The foods provided in this diet will be closely aligned with the NHANES "What we eat in America" report.
  Arms: NHANES Diet Plan

SUMMARY:
To determine if consumption of different diet plans that both are nutritionally-adequate and provide energy to maintain body weight, alters fasting insulin concentrations, shifts other common clinical markers of metabolic disease risk, and affects metabolomic profiles that reflect glucose, lipid, and amino acid metabolism.

DETAILED DESCRIPTION:
Western Human Nutrition Research Center (WHNRC) scientists have observed rapid and substantial improvements in metabolic health indices in non-diabetic obese persons who undergo a weight-maintenance diet including prepared meals that were aligned with current dietary recommendations, including those of the Institute of Medicine and the United States Department of Agriculture (USDA) and Department of Health and Human Services (DHHS) Dietary Guidelines for Americans. For instance, marked reductions and often normalization of hyperinsulinemia were observed within days of provision of a controlled nutrient-dense high quality diet, and LDL was reduced by 20-30% or more within 2 weeks or possibly earlier. This indicates that change in diet alone would benefit many at-risk persons with respect to normalizing metabolic parameters and disease risk markers. Yet, surprisingly little formal research has focused on how a high quality, weight maintaining diet impacts health over a short-term period in at-risk individuals. The overall objective of this study is to determine if a nutrient-adequate diet closely aligned with food group recommendations set in the 2010 Dietary Guidelines for Americans elicits a superior metabolic profile in persons at-risk for metabolic disease, compared to a nutrient-adequate containing foods closely aligned with the National Health and Nutrition Examination Survey (NHANES) "What We Eat In America" report. Further, the investigation will include effect modification of stress-related cortisol measures on change in cardiometabolic risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal by self-report
* Body Mass Index 25-39.9 kg/m2
* Fasting glucose ≥100 and <126 mg/dL and/or
* Oral Glucose Tolerance Test (OGTT) 2-hour glucose ≥140 and <199 mg/dL and/or
* Quantitative insulin sensitivity check index (QUICKI) score <0.315 and/or
* Homeostasis Model Assessment (HOMA) >3.67, or log HOMA >0.085 and/or
* Glycated Hemoglobin HbA1c ≥5.7 and <6.5fasting glucose ≥100 and <126 mg/dL and/or
* Fasting triglyceride concentrations >150 mg/dL and/or
* LDL cholesterol >100 mg/dL and/or
* HDL cholesterol <40 mg/dL.

Exclusion Criteria:

* BMI <25 and >39.9 kg/m2
* Presence of any metabolic diseases, by self-report
* Gastrointestinal disorders by self-report
* Presence of cancer or other serious chronic disease by self-report
* Current use of prescribed or over the counter weight loss medications
* Pregnant
* Lactating
* Current use of tobacco
* Moderate or strenuous physical activity >30 min/day, 5 or more days per week
* Weight change >5% of body weight during the previous 6 months
* Dietary restrictions that would interfere with consuming the intervention foods

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2014-12-16 (Actual); Primary Completion 2017-03-30 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
Change in Fasting Insulin Concentrations | Weeks 1, 3, and 9
  Additional indicators of glucose-insulin sensitivity will be assessed including the Quantitative Insulin Sensitivity Check Index (QUICKI) score, Homeostasis Model Assessment (HOMA), and Matsuda Index

SECONDARY OUTCOMES:
Change in Lipid Profile | Weeks 1, 3, and 9
  fasting triglyceride concentrations, LDL cholesterol, HDL cholesterol will be measured in serum as a composite measurement

OTHER OUTCOMES:
Change in Metabolomic Profile | Weeks 1,3, and 9
  Endocannabinoids, Bile Acids, Amino Acids, Acyl Carnitines, Non-Esterified Fatty Acids, Oxylipins, Corticoids, Nitrate/Nitrite, and Tissue Lipid Profile will be measured in plasma, erythrocytes, and sebaceous secretions as a composite measurement.
Change in Immunological Markers | Weeks 1 and 9
  Immunologic markers such as tumor necrosis factor-α, Interleukin-β, Interleukin-6, Interferon-γ, Interleukin-13, Interleukin-17A, Interleukin-10 will be measured in plasma and whole cell preparations as a composite measurement.
Bio-Behavioral responses to diet intervention | Weeks 1 and 9
  Stress Reactivity, Allostatic Load, Autonomic Nervous System Output, and Cognitive Function will be recorded as a composite measurement.
Change in responses to Behavioral questionnaires | Weeks 1, 3, and 9
  Appetite, Food Preference, Diet Bias will be measured and reported as a composite measurement.
Change in Taste preference threshold | Weeks 1 and 9
  Sweet, salty, and bitter taste sensitivity will be evaluated using the three-alternative-forced choice method for determining recognition taste thresholds
Change in intestinal microbiota | weeks 1, 3, 5 and 9
  Assays will be performed on fecal samples to determine DNA representing the colonic microbiota, amount of organic acids and other metabolites of fermentation.
Change in usual physical activity | weeks 1, 3, and 9
  Usual physical activity will be measured by accelerometer worn for 7 days
Change in body composition | weeks 1 and 9
  Body composition (total body fat) will be measured by dual energy x-ray absorptiometry (DXA)
Change in vascular function | weeks 1 and 9
  Vascular function assessment of peripheral arterial tone (PAT) measurement conducted at resting conditions and after a reactive hyperemia
Change in Framingham Risk Score | weeks 1, 3 and 9
  Calculated Framingham 10-year cardiovascular disease risk score
Change in vascular age score | weeks 1, 3 and 9
  Calculated vascular age score
Change in metabolic rate | weeks 1, 3, and 9
  Respiratory gas exchange measurements (oxygen consumption and carbon dioxide production) will be measured in response to a test meal
Change in breath volatile gases | weeks 1, 3, and 9
  Alveolar air (breath) samples will be analyzed for hydrogen and methane, products produced by bacterial fermentation of carbohydrates in the gastrointestinal tract
Usual diet | week 1
  Usual diet will be measured once by food frequency questionnaire and 24 hour recall methodology
Change in post-translational glycosylation of select serum proteins (glycoproteome) | weeks 1, 3 and 9
  Serum circulating protein concentrations and their glycovariant distributions measured by Ultra High Pressure Liquid Chromatography - Mass Spectrometry (UHPLC-MS). Proteins selected based on their association to chronic metabolic disease, such as angiotensinogen, fibronectin, kininogen, kallikrein, apolipoprotein CIII, fetuin and vitronectin.
Change in Trimethylamine Oxide (TMAO) | weeks 1, 3 and 9
  Fasting serum level of TMAO measured by liquid chromatography mass spectrometry (LCMS)
Change in choline | weeks 1, 3 and 9
  Fasting serum level of choline measured by liquid chromatography mass spectrometry (LCMS)
Change in carnitine | weeks 1, 3 and 9
  Fasting serum level of carnitine measured by liquid chromatography mass spectrometry (LCMS)
Change in betaine | weeks 1, 3 and 9
  Fasting serum level of betaine measured by liquid chromatography mass spectrometry (LCMS)
Change in creatinine | weeks 1, 3 and 9
  Fasting serum level of creatinine measured by liquid chromatography mass spectrometry (LCMS)
Fasting urinary cortisol | weeks 1 and 9
  Cortisol was measured in 12-hour overnight urine samples collected prior to eating
Baseline and change in diurnal salivary cortisol | weeks 1 and 9; at nighttime before going to sleep and upon waking
  Cortisol was measured in saliva samples collected using a cotton swab (Salivette)
Baseline and change in salivary cortisol response to a meal | weeks 1 and 9; at 60, 90, and 120 minutes after the initiation of a meal
  Cortisol was measured in saliva samples collected using a cotton swab (Salivette)
Baseline and change in salivary cortisol response to stress | weeks 1 and 9; at 30, 60, 90, and 120 minutes after the start of a stress test
  Cortisol was measured in saliva samples collected using a cotton swab (Salivette)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy L Keim, PhD, Principal Investigator — USDA, Western Human Nutrition Research Center
Locations (2):
- United States (2):
  - Western Human Nutrition Research Center, Davis, California
  - Clinical Translational Science Center, Sacramento, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Krishnan S, Freytag T, Jiang X, Schuster GU, Woodhouse LR, Keim NL, Stephensen CB. Effect of a diet based on the dietary guidelines for americans on inflammation markers in women at risk for cardiometabolic disease: results of a randomized, controlled trial. BMC Nutr. 2022 Dec 27;8(1):157. doi: 10.1186/s40795-022-00647-z. PMID 36575541
- [Derived] Soltani H, Keim NL, Laugero KD. Waking Salivary Cortisol Associated with Magnitude of Cholesterol Reduction in Women Fed a Healthy Whole-Food Diet for 8 Weeks. Curr Dev Nutr. 2022 May 3;6(5):nzac083. doi: 10.1093/cdn/nzac083. eCollection 2022 May. PMID 35669046
- [Derived] Newman JW, Krishnan S, Borkowski K, Adams SH, Stephensen CB, Keim NL. Assessing Insulin Sensitivity and Postprandial Triglyceridemic Response Phenotypes With a Mixed Macronutrient Tolerance Test. Front Nutr. 2022 May 11;9:877696. doi: 10.3389/fnut.2022.877696. eCollection 2022. PMID 35634390
- [Derived] Richardson CE, Krishnan S, Gray IJ, Keim NL, Newman JW. The Omega-3 Index Response to an 8 Week Randomized Intervention Containing Three Fatty Fish Meals Per Week Is Influenced by Adiposity in Overweight to Obese Women. Front Nutr. 2022 Feb 4;9:810003. doi: 10.3389/fnut.2022.810003. eCollection 2022. PMID 35187036
- [Derived] Krishnan S, Gertz ER, Adams SH, Newman JW, Pedersen TL, Keim NL, Bennett BJ. Effects of a diet based on the Dietary Guidelines on vascular health and TMAO in women with cardiometabolic risk factors. Nutr Metab Cardiovasc Dis. 2022 Jan;32(1):210-219. doi: 10.1016/j.numecd.2021.09.013. Epub 2021 Sep 20. PMID 34895998
- [Derived] Artegoitia VM, Krishnan S, Bonnel EL, Stephensen CB, Keim NL, Newman JW. Healthy eating index patterns in adults by sex and age predict cardiometabolic risk factors in a cross-sectional study. BMC Nutr. 2021 Jun 22;7(1):30. doi: 10.1186/s40795-021-00432-4. PMID 34154665
- [Derived] Kim T, Xie Y, Li Q, Artegoitia VM, Lebrilla CB, Keim NL, Adams SH, Krishnan S. Diet affects glycosylation of serum proteins in women at risk for cardiometabolic disease. Eur J Nutr. 2021 Oct;60(7):3727-3741. doi: 10.1007/s00394-021-02539-7. Epub 2021 Mar 26. PMID 33770218
- [Derived] Krishnan S, Lee F, Burnett DJ, Kan A, Bonnel EL, Allen LH, Adams SH, Keim NL. Challenges in Designing and Delivering Diets and Assessing Adherence: A Randomized Controlled Trial Evaluating the 2010 Dietary Guidelines for Americans. Curr Dev Nutr. 2020 Feb 13;4(3):nzaa022. doi: 10.1093/cdn/nzaa022. eCollection 2020 Mar. PMID 32190808
- [Derived] Krishnan S, Adams SH, Allen LH, Laugero KD, Newman JW, Stephensen CB, Burnett DJ, Witbracht M, Welch LC, Que ES, Keim NL. A randomized controlled-feeding trial based on the Dietary Guidelines for Americans on cardiometabolic health indexes. Am J Clin Nutr. 2018 Aug 1;108(2):266-278. doi: 10.1093/ajcn/nqy113. PMID 30101333
- See also: USDA Western Human Nutrition Research Center — http://www.ars.usda.gov/main/docs.htm?docid=11240